CLINICAL TRIAL: NCT02013037
Title: The De-novo Use of Eculizumab Alongside Conventional Therapy in Presensitized Patients Receiving Cardiac Transplantation: An Open-Label, Investigator-Initiated Pilot Trial: [The DUET Cardiac Trial]
Brief Title: The De-novo Use of Eculizumab in Presensitized Patients Receiving Cardiac Transplantation
Acronym: DUET
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Collaborators: Alexion Pharmaceuticals, Inc. (Industry)
Responsible Party: Principal Investigator, Jignesh Patel, MD, PhD, Medical Director of Heart Transplant Program, Cedars Sinai Heart Institute, Cedars-Sinai Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSR 205237; Pro00028970 (Other: Cedars-Sinai Medical Ctr. IRB)
Record Dates: First submitted 2013-12-11; First posted 2013-12-17 (Estimated); Results first posted 2021-05-03 (Actual); Last update posted 2021-05-03 (Actual); Status verified 2021-04

CONDITIONS: Antibody-mediated Rejection; Hyperacute Rejection of Cardiac Transplant; Left Ventricular Dysfunction; Cardiac Allograft Vasculopathy; Heart Graft Dysfunction
Keywords: cardiac transplantation; immunosuppression; acute cellular rejection; antibody mediated rejection; sensitization; antibody production in cardiac patients; panel reactive antibodies; desensitization strategies in heart transplant patients; complement activation; complement c3d and c4d deposition; terminal complement inhibition; complement C5 binding; Eculizumab; monoclonal antibody; donor specific antibodies
MeSH Terms: conditions — Ventricular Dysfunction, Left; Complement Component 3 Deficiency, Autosomal Recessive | interventions — eculizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Eculizumab (Experimental): Administration of Eculizumab to heart transplant recipients at Cedars Sinai Medical Center with a panel reactive antibody (PRA) ≥ 70%, for the prevention of antibody-mediated rejection.
  Interventions: Drug: Eculizumab

INTERVENTIONS:
Drug: Eculizumab — At the time of transplantation, 1200mg of Eculizumab will be administered via a 35 minute IV infusion, followed by thymoglobulin 1.5 mg/kg intravenous piggyback (IVPB). The administration of thymoglobulin will be repeated (if blood counts permit) for a total of five doses.
  On Day 1 post-transplant, 900 mg of Eculizumab will be given via an IV infusion.
  On Day 5 post-transplant, intravenous immunoglobulin (IVIG) 1 gram/kg will be administered daily for two consecutive days.
  On post-transplant days 7, 14, and 21 (+/- 2 days) 900mg of Eculizumab will be given via an IV infusion at each scheduled visit.
  On post-transplant days 28, 42, and 56 (+/- 2 days) 1200 mg of Eculizumab will be given via an IV infusion at each scheduled visit.
  Other Names: Soliris

SUMMARY:
All individuals who receive a heart transplant are at risk for developing antibody-mediated rejection (AMR). An antibody is a protein produced by the body's immune system when it detects a foreign substance, called an antigen. The mechanism of an antibody is to attack an antigen. In antibody mediated rejection, antibodies will attack the transplanted heart, causing injury to the heart. The purpose of this investigation is to determine if a study drug, called eculizumab (Soliris), is safe to use in heart transplant recipients, and determine if it reduces risk of antibody-mediated rejection.

DETAILED DESCRIPTION:
The growing proportion of sensitized cardiac recipients presents an additional challenge to the transplant practitioner attempting to minimize the occurrence of antibody mediated rejection (AMR). Patients pre-exposed or "sensitized" to antigen exposing events (i.e.: blood transfusions, multiple pregnancies, prior organ transplantations, ventricular support devices) are more likely to both possess preformed and develop de-novo antibodies. Sensitized patients with panel reactive antibodies > 25% are at risk for increased risk of rejection, development of cardiac allograft vasculopathy and increased mortality after heart transplantation.

A central component of antibody-mediated cell injury is complement activation. The inhibition of terminal complement activation may be the missing link to decreasing possibly both complement-mediated AMR and cellular rejection (CR) by inhibiting both the inflammatory effects of both circulating antibodies and cytokine induced cell death.

Eculizumab is a monoclonal antibody that specifically binds to complement protein C5 with high affinity, thereby inhibiting its cleavage to C5a and C5b and preventing the generation of the terminal complement complex C5b-9. By this mechanism, eculizumab (Soliris®) inhibits terminal complement mediated intravascular hemolysis in paroxysmal nocturnal hemoglobinuria patients.

This study is a non-randomized, open-label, investigator-initiated safety and efficacy trial investigating the de-novo use of eculizumab alongside conventional therapy to prevent antibody mediated rejection. The duration of the study will include an open enrollment period and at least 12 months of follow-up (post-transplant). We will consent up to 45 eligible patients, highly "sensitized", with a panel reactive antibody score greater than 70%, who are not previously or currently enrolled in another ongoing trial. Of these 45 participants, up to 20 of these patients will be treated with eculizumab (Solaris), the study drug. The use of eculizumab will be un-blinded to all study and research practitioner participants.

ELIGIBILITY:
Inclusion Criteria:

* Patient is ≥ 18 years of age.
* Patient has a panel reactive antibody (PRA) ≥ 70% at any time prior to screening.
* Patient is considered compliant and intends to be available for a minimum follow-up study period of 1 year.
* Patient must be vaccinated against Neisseria meningitides at least 2 weeks prior to receiving treatment therapy or receive appropriate antibiotic prophylaxis for the duration of eculizumab treatment if timely vaccination could not be achieved prior to transplantation.
* Voluntary written informed consent must be obtained before performance of any study-related procedure not considered routine medical care, with the understanding that consent may be withdrawn by the subject at any time without prejudice to future medical care.
* Female subject is either post-menopausal or surgically sterilized or willing to use two acceptable methods of birth control (i.e., a hormonal contraceptive, intra-uterine device, diaphragm with spermicide, condom with spermicide, or abstinence) for the duration of the study and for up to 2 months after the last dose of study medication.

Exclusion Criteria:

* Donor or recipient age is < 18 years or > 75 years.
* Cold ischemia time is > 6 hours.
* Current clinical, radiographic, or laboratory evidence of active or latent tuberculosis (TB), as determined by local standard of care.
* History of active TB within the last 2 years, even if treated.
* History of active TB greater than 2 years ago, unless there is documentation of adequate treatment according to locally accepted clinical practice.

(Note: Patients at risk of TB reactivation preclude administration of conventional immunosuppression, as determined by the study investigator and based upon appropriate evaluation).

* Receipt of desensitization treatment with rituximab less than 2 weeks prior to therapy and cluster of differentiation antigen 20 (CD20) count >2%.
* Receipt of a live vaccine within 4 weeks prior to study entry.
* Patients with current or recent severe systemic infections within the 2 weeks prior to transplantation.
* Prior history of splenectomy.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2012-11; Primary Completion 2019-12-30 (Actual); Study Completion 2020-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jignesh Patel, M.D., Ph.D., Principal Investigator — Cedars Sinai Medical Center and Heart Institute
Locations (1):
- Cedars Sinai Medical Center, Heart Institute, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that supports the results of the study after deidentification and in accordance with Cedars Sinai data sharing agreements.
Supporting Information: Study Protocol, SAP
Time Frame: Data will be available following publication and ending 3 years following article publication.
Access Criteria: Data will be available to investigators whose proposed used of the data has been approved by Cedars Sinai IRB.

REFERENCES:
- [Background] Kfoury AG, Hammond ME, Snow GL, Drakos SG, Stehlik J, Fisher PW, Reid BB, Everitt MD, Bader FM, Renlund DG. Cardiovascular mortality among heart transplant recipients with asymptomatic antibody-mediated or stable mixed cellular and antibody-mediated rejection. J Heart Lung Transplant. 2009 Aug;28(8):781-4. doi: 10.1016/j.healun.2009.04.035. PMID 19632573
- [Background] Uber WE, Self SE, Van Bakel AB, Pereira NL. Acute antibody-mediated rejection following heart transplantation. Am J Transplant. 2007 Sep;7(9):2064-74. doi: 10.1111/j.1600-6143.2007.01900.x. Epub 2007 Jul 5. PMID 17614978
- [Background] Wu GW, Kobashigawa JA, Fishbein MC, Patel JK, Kittleson MM, Reed EF, Kiyosaki KK, Ardehali A. Asymptomatic antibody-mediated rejection after heart transplantation predicts poor outcomes. J Heart Lung Transplant. 2009 May;28(5):417-22. doi: 10.1016/j.healun.2009.01.015. Epub 2009 Mar 14. PMID 19416767
- [Background] Michaels PJ, Espejo ML, Kobashigawa J, Alejos JC, Burch C, Takemoto S, Reed EF, Fishbein MC. Humoral rejection in cardiac transplantation: risk factors, hemodynamic consequences and relationship to transplant coronary artery disease. J Heart Lung Transplant. 2003 Jan;22(1):58-69. doi: 10.1016/s1053-2498(02)00472-2. PMID 12531414
- [Background] Stegall MD, Diwan T, Raghavaiah S, Cornell LD, Burns J, Dean PG, Cosio FG, Gandhi MJ, Kremers W, Gloor JM. Terminal complement inhibition decreases antibody-mediated rejection in sensitized renal transplant recipients. Am J Transplant. 2011 Nov;11(11):2405-13. doi: 10.1111/j.1600-6143.2011.03757.x. Epub 2011 Sep 22. PMID 21942930
- [Background] Nwakanma LU, Williams JA, Weiss ES, Russell SD, Baumgartner WA, Conte JV. Influence of pretransplant panel-reactive antibody on outcomes in 8,160 heart transplant recipients in recent era. Ann Thorac Surg. 2007 Nov;84(5):1556-62; discussion 1562-3. doi: 10.1016/j.athoracsur.2007.05.095. PMID 17954062
- [Background] Kobashigawa J, Crespo-Leiro MG, Ensminger SM, Reichenspurner H, Angelini A, Berry G, Burke M, Czer L, Hiemann N, Kfoury AG, Mancini D, Mohacsi P, Patel J, Pereira N, Platt JL, Reed EF, Reinsmoen N, Rodriguez ER, Rose ML, Russell SD, Starling R, Suciu-Foca N, Tallaj J, Taylor DO, Van Bakel A, West L, Zeevi A, Zuckermann A; Consensus Conference Participants. Report from a consensus conference on antibody-mediated rejection in heart transplantation. J Heart Lung Transplant. 2011 Mar;30(3):252-69. doi: 10.1016/j.healun.2010.11.003. PMID 21300295
- [Background] Berry GJ, Angelini A, Burke MM, Bruneval P, Fishbein MC, Hammond E, Miller D, Neil D, Revelo MP, Rodriguez ER, Stewart S, Tan CD, Winters GL, Kobashigawa J, Mehra MR. The ISHLT working formulation for pathologic diagnosis of antibody-mediated rejection in heart transplantation: evolution and current status (2005-2011). J Heart Lung Transplant. 2011 Jun;30(6):601-11. doi: 10.1016/j.healun.2011.02.015. No abstract available. PMID 21555100
- [Background] Locke JE, Magro CM, Singer AL, Segev DL, Haas M, Hillel AT, King KE, Kraus E, Lees LM, Melancon JK, Stewart ZA, Warren DS, Zachary AA, Montgomery RA. The use of antibody to complement protein C5 for salvage treatment of severe antibody-mediated rejection. Am J Transplant. 2009 Jan;9(1):231-5. doi: 10.1111/j.1600-6143.2008.02451.x. Epub 2008 Oct 31. PMID 18976298
- [Background] Wang H, Arp J, Liu W, Faas SJ, Jiang J, Gies DR, Ramcharran S, Garcia B, Zhong R, Rother RP. Inhibition of terminal complement components in presensitized transplant recipients prevents antibody-mediated rejection leading to long-term graft survival and accommodation. J Immunol. 2007 Oct 1;179(7):4451-63. doi: 10.4049/jimmunol.179.7.4451. PMID 17878341
- [Background] Thomas TC, Rollins SA, Rother RP, Giannoni MA, Hartman SL, Elliott EA, Nye SH, Matis LA, Squinto SP, Evans MJ. Inhibition of complement activity by humanized anti-C5 antibody and single-chain Fv. Mol Immunol. 1996 Dec;33(17-18):1389-401. doi: 10.1016/s0161-5890(96)00078-8. PMID 9171898
- [Background] Rinder CS, Rinder HM, Smith BR, Fitch JC, Smith MJ, Tracey JB, Matis LA, Squinto SP, Rollins SA. Blockade of C5a and C5b-9 generation inhibits leukocyte and platelet activation during extracorporeal circulation. J Clin Invest. 1995 Sep;96(3):1564-72. doi: 10.1172/JCI118195. PMID 7657827
- [Derived] Coutance G, Kobashigawa JA, Kransdorf E, Loupy A, Desire E, Kittleson M, Patel JK. Intermediate-term outcomes of complement inhibition for prevention of antibody-mediated rejection in immunologically high-risk heart allograft recipients. J Heart Lung Transplant. 2023 Oct;42(10):1464-1468. doi: 10.1016/j.healun.2023.05.005. Epub 2023 May 12. PMID 37182818
- [Derived] Patel JK, Coutance G, Loupy A, Dilibero D, Hamilton M, Kittleson M, Kransdorf E, Azarbal B, Seguchi O, Zhang X, Chang D, Geft D, Czer L, Varnous S, Kobashigawa JA. Complement inhibition for prevention of antibody-mediated rejection in immunologically high-risk heart allograft recipients. Am J Transplant. 2021 Jul;21(7):2479-2488. doi: 10.1111/ajt.16420. Epub 2021 Feb 11. PMID 33251691

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled following written informed consent for a protocol approved by the Institutional Review Board of Cedars-Sinai Medical Center (NCT02013037).The duration of the study included an open enrollment period and at least 12 months of post-transplant follow-up. All patients worked up for a heart transplant at the Heart Institute at Cedars-Sinai Medical Center (CSMC) with a panel reactive antibody (PRA) ≥ 70% at any time prior to screening.
Pre-assignment Details: The trial enrolled a total of 36 sensitized participants age ≥ 18 years with a panel reactive antibody ≥70% at any time prior to study screening. Participants were included in the eculizumab treatment group if at least one donor specific antibody at MFI≥5000 was crossed but with negative prospective complement-dependent cytotoxicity crossmatch. 16 enrolled patients did not receive eculizumab.
Period: Overall Study
Arm/Group | Eculizumab
Started | 36
Completed | 20
Not Completed | 16
Not completed — Death | 6
Not completed — Withdrawal by Subject | 1
Not completed — Awaiting Transplantation | 7
Not completed — Transplanted without DSA | 2

BASELINE CHARACTERISTICS:
Population: The trial enrolled a total of 36 sensitized participants age ≥ 18 years with a panel reactive antibody (PRA) ≥70% at any time prior to study screening. Participants were included in the eculizumab treatment group if at least one DSA at MFI≥ 5000 was crossed but with negative prospective complement-dependent cytotoxicity (CDC) crossmatch. The eculizumab group consisted of 20 consecutive recipients transplanted between June 2, 2013 and July 31, 2018.
Arm/Group | Eculizumab
Number analyzed (Participants) | 20
Age, Continuous [Median (Full Range); unit: years] | 53.3 [44 to 60.2]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 4
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Non-Caucasian | 7
Region of Enrollment [Number; unit: participants]
  United States | 20
Non ischemic heart failure [Count of Participants; unit: Participants] | 15
Time on waiting list [Median (Full Range); unit: Days] | 129 [46 to 198]
Long term mechanical circulatory support (MCS) or extra-corporeal membrane oxygena at transplant [Count of Participants; unit: Participants] | 10
Combined transplantation [Count of Participants; unit: Participants] | 2
Retransplantation [Count of Participants; unit: Participants] | 5
Prior blood transfusion [Count of Participants; unit: Participants] | 8
Prior pregnancy (women) [Count of Participants; unit: Participants] — Population: The analysis population includes only the number of women (16)
  Participants
    number analyzed (Participants) | 16
    (all) | 14
Pre-transplant diabetes [Count of Participants; unit: Participants] | 7
Pre-transplant hypertension [Count of Participants; unit: Participants] | 8
Serum creatinine [Median (Full Range); unit: mg/dL] | 1.35 [1 to 1.65]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants of Pathologic Antibody-Mediated Rejection and Left Ventricular Dysfunction
Description: The efficacy of Eculizumab will be assessed by a composite endpoint of:
  1. the incidence of pathologic AMR with a Grade ≥ 2
  2. the incidence of left ventricular dysfunction, as defined by a left ventricular ejection fraction (LVEF) ≤ 40% or a decrease of >15% from baseline prior to the initiation of Eculizumab treatment.
Time Frame: up to 26 weeks post heart transplant
Measure: Count of Participants; unit: Participants
Groups:
- Eculizumab: Administration of Eculizumab to heart transplant recipients at Cedars Sinai Medical Center with a panel reactive antibody (PRA) ≥ 70%, for the prevention of antibody-mediated rejection.
  Eculizumab: At the time of transplantation, 1200mg of Eculizumab will be administered via a 35 minute IV infusion, followed by thymoglobulin 1.5 mg/kg intravenous piggyback (IVPB). The administration of thymoglobulin will be repeated (if blood counts permit) for a total of five doses.
  On Day 1 post-transplant, 900 mg of Eculizumab will be given via an IV infusion.
  On Day 5 post-transplant, intravenous immunoglobulin (IVIG) 1 gram/kg will be administered daily for two consecutive days.
  On post-transplant days 7, 14, and 21 (+/- 2 days) 900mg of Eculizumab will be given via an IV infusion at each scheduled visit.
  On post-transplant days 28, 42, and 56 (+/- 2 days) 1200 mg of Eculizumab will be given via an IV infusion at each scheduled visit.
Arm/Group | Eculizumab
Number analyzed (Participants) | 20
Participants | 4

2. Secondary Outcome: Patient Survival at 12 Months Post Heart Transplantation
Description: The study will assess overall survival at 12 months following heart transplantation.
Time Frame: 1 year post heart transplant
Population: 20 participants were included in the Eculizumab study
Measure: Count of Participants; unit: Participants
Arm/Group | Eculizumab
Number analyzed (Participants) | 20
Participants | 18

3. Secondary Outcome: Number of Participants With Hemodynamic Compromise at 6 Months Post Transplant
Description: The incidence of patient hemodynamic compromise will be assessed at 6 months post transplant, as defined by any one of the following:
  1. a 20% decrease in LVEF from baseline
  2. a LVEF < 40%
  3. a 25% decrease in cardiac index from baseline
  4. a cardiac index < 2.0
  5. the need for inotropic support
Time Frame: 6 months post heart transplant
Population: 20 participants were included in the Eculizumab study
Measure: Count of Participants; unit: Participants
Arm/Group | Eculizumab
Number analyzed (Participants) | 20
Participants | 0

4. Secondary Outcome: Number of Participants With Hemodynamic Compromise at 1 Year Post Transplant
Description: The incidence of patient hemodynamic compromise will be assessed at one year post transplant, as defined by any one of the following:
  1. a 20% decrease in LVEF from baseline
  2. a LVEF < 40%
  3. a 25% decrease in cardiac index from baseline
  4. a cardiac index < 2.0
  5. the need for inotropic support
Time Frame: 1 year post heart transplant
Population: 20 participants participated in the eculizumab study
Measure: Count of Participants; unit: Participants
Arm/Group | Eculizumab
Number analyzed (Participants) | 20
Participants | 0

5. Secondary Outcome: Number of Participants With Antibody Mediated Rejection (AMR)
Description: The study assessed the number of patients who develop AMR as well as the total number of episodes of AMR.
Time Frame: up to 1 year post heart transplant
Population: 20 participants were treated in the eculizumab study
Measure: Count of Participants; unit: Participants
Arm/Group | Eculizumab
Number analyzed (Participants) | 20
Participants | 6

6. Secondary Outcome: Number of Participants With of Acute Cellular Rejection (ACR)
Description: The study assessed the number of participants with of Acute Cellular Rejection (ACR)
Time Frame: up to 1 year post heart transplant
Population: 20 participants were treated in the eculizumab study
Measure: Count of Participants; unit: Participants
Arm/Group | Eculizumab
Number analyzed (Participants) | 20
Participants | 0

7. Secondary Outcome: Development of Cardiac Allograft Vasculopathy (CAV) by Intravascular Ultrasound (IVUS)
Description: Development of cardiac allograft vasculopathy at 1 year determined by intravascular ultrasound defined as change in site-matched maximal intimal thickness ≥ 0.5mm from baseline to 1 year.
Time Frame: up to 1 year post heart transplant
Population: 20 enrolled patients were treated on the study
Measure: Count of Participants; unit: Participants
Arm/Group | Eculizumab
Number analyzed (Participants) | 20
Participants | 1

8. Secondary Outcome: Number of Participants With Evolution of DSA: Donor Specific Antibody Post Transplantation
Description: Number of Participants who develop de novo donor specific antibody (DSA) in the first year following transplantation was determined.
Time Frame: Up to 1 year post transplant
Population: 20 enrolled patients were treated on the study
Measure: Count of Participants; unit: Participants
Arm/Group | Eculizumab
Number analyzed (Participants) | 20
Participants | 5

ADVERSE EVENTS:
Time Frame: 1 year post transplant
Groups:
- Eculizumab: Administration of Eculizumab to heart transplant recipients at Cedars Sinai Medical Center with a panel reactive antibody (PRA) ≥ 70%, for the prevention of antibody-mediated rejection.
  Eculizumab: At the time of transplantation, 1200mg of Eculizumab will be administered via a 35 minute IV infusion, followed by thymoglobulin 1.5 mg/kg intravenous piggyback (IVPB). The administration of thymoglobulin will be repeated (if blood counts permit) for a total of five doses.
  On Day 1 post-transplant, 900 mg of Eculizumab will be given via an IV infusion.
  On Day 5 post-transplant, intravenous immunoglobulin (IVIG) 1 gram/kg will be administered daily for two consecutive days.
  On post-transplant days 7, 14, and 21 (+/- 2 days) 900mg of Eculizumab will be given via an IV infusion at each scheduled visit.
  On post-transplant days 28, 42, and 56 (+/- 2 days) 1200 mg of Eculizumab will be given via an IV infusion at each scheduled visit.
  2 deaths were reported in participants who received eculizumab. There were 6 deaths in participants who did not complete the study and did not receive eculizumab.
Arm/Group | Eculizumab
All-Cause Mortality (participants affected / at risk) | 8/36
Serious Adverse Events (participants affected / at risk) | 13/36
Other Adverse Events (participants affected / at risk) | 0/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Eculizumab (N=36)
Viral infections (Infections and infestations) | 6 (6)
Bacterial Infections (Infections and infestations) | 7 (8)
Fungal infections (Infections and infestations) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan: Study Protocol including Statistical Analysis Plan (2015-07-09): https://cdn.clinicaltrials.gov/large-docs/37/NCT02013037/Prot_SAP_000.pdf